CLINICAL TRIAL: NCT00872703
Title: Does Normal Brain Imaging Predict Normal Neurodevelopmental Outcome in Fetuses With Proven Cytomegalovirus Infection?
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Sheba Medical Center (Other Government); Tel Aviv Medical Center (Other)
Responsible Party: Gustavo Malinger, MD, Director OB-GYN Ultrasound Unit
Other Study IDs: SR-907
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: CMV; Prenatal Diagnosis; Ultrasound; MRI
Keywords: CMV; Prenatal Diagnosis; Ultrasound; MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Cytomegalovirus (CMV) is the largest member of the virus family Herpesviridae that infects almost all humans at some point in their lives (Ross, 2004). Congenital CMV infection is most likely to occur when the mother experiences a primary infection during pregnancy, and it is much less common in cases of reactivation of the disease or infection by a different CMV strain (Boppana 1999, Endres 2001). The prevalence of congenital CMV infection varies between 0.15-2.2% (Ross 2004, Ross 2006, Malm 2007). While most infants born with congenital CMV infection are asymptomatic, 10 to 15% show clinical findings at birth (Ross 2004).

It is generally agreed that congenital CMV infection, whether it is symptomatic or not, is a major risk factor for perceptual deficits. However, its influence on children's future neuropsychological functioning is less well established. Symptomatic congenital CMV infection is a major risk factor for poor developmental outcome (Williamson 1982, Kylat 2006, Dollard 2007), but the available data regarding neuropsychological outcome for asymptomatic children is extremely diverse (Conboy 1986, Ivarson 1997, Kashdan 1998, Temple 2000, Zhang 2007).

We evaluated the neuropsychological outcome of children with congenital cytomegalovirus (CMV) infection and normal consecutive fetal neurosonographic examinations and determined whether Magnetic Resonance Imaging (MRI) provided additional information in these cases.

ELIGIBILITY:
Inclusion Criteria:

* CMV PCR positive in the amniotic fluid

Exclusion Criteria:

* US abnormal findings during fetal life

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children of woman with CMV proved intrauterine infections
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
neuropsychological outcome | 1-7 years

CONTACTS AND LOCATIONS:
Locations (1):
- E. Wolfson Medical Center, Holon, Israel